CLINICAL TRIAL: NCT04954469
Title: B-pVAC-SARS-CoV-2: Phase I/II Multicenter Safety and Immunogenicity Trial of Multi-peptide Vaccination to Prevent COVID-19 Infection in Adults With Bcell/ Antibody Deficiency
Brief Title: B-pVAC-SARS-CoV-2: Study to Prevent COVID-19 Infection in Adults With Bcell/ Antibody Deficiency
Acronym: B-pVAC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-pVAC-SARS-CoV-2
Record Dates: First submitted 2021-07-05; First posted 2021-07-08 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2022-11

CONDITIONS: Immune Deficiency Disease
MeSH Terms: conditions — Immune Deficiency Disease | interventions — COVAC-1 COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Phase I:
  Part I: 14 patients not infected with SARS-CoV-2 will receive an open-label 500 μl subcutaneous injection via needle and syringe of the study IMP (CoVAC-1).
  Part II (optional): If there is an insufficient immune response measured by IFN-γ ELISpot in Part I of Phase I on day 28, an additional Part (Part II) of Phase I will start enrollment of 14 subjects receiving two open-label 500 μl subcutaneous injection via needle and syringe of the study IMP (CoVac-1) on d1 and d42.
  Phase II (after an amendment to the protocol):
  40 subjects will receive an open-label 500 μl subcutaneous injection via needle and syringe of the study IMP (CoVac-1) on d1 and, depending on the data collected in Phase I, a econd vaccination on d42 if necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CoVAC-1 Vaccine (Experimental): Peptide vaccination should be started as soon as possible after the screening visit. Or in case of two vaccinations: Peptide vaccination should be started as soon as possible after the screening visit (V1) and on day 42 (V5)
  Interventions: Biological: CoVAC-1

INTERVENTIONS:
Biological: CoVAC-1 — Peptide vaccination should be started as soon as possible after the screening visit.

SUMMARY:
The indication of this study is To evaluate the safety and immunogenicity of a SARSCoV- 2-derived multi-peptide vaccine in combination with the TLR1/2 ligand XS15 in adults with congenital or acquired B-cell/antibody deficiency

DETAILED DESCRIPTION:
Multicenter Phase I-II clinical trial

Phase I:

Part I: 14-patients will receive an open-label 500 μl subcutaneous injection via needle and syringe of the study IMP (CoVac-1). 28 days following vaccination of the

1th patient, there will be an interim analysis of safety and immunogenicity and a review by the data safety monitoring board (DSMB) before proceeding to Phase II Definition of sufficient immunogenicity after one dose of vaccination: T cell response to at least one CoVAC-1 vaccine peptide on day28 in ≥80% of study patients, with proven general ability to mount antigen-specific T cell responses (detection of T cell responses to EBV/CMV control peptides) assessed by Interferon gamma (IFN-γ) ELISpot.

* The time point (day28) for the assessment of CoVac-1 induced T cell responses was selected based on the results of the ongoing P-pVAC-SARS-CoV-2 study, where CoVac-1-induced SARS-CoV-2 T cell responses were observed in 100% of study subjects at day28.
* The threshold of 80% was introduced after considering recent findings about cancer patients with hematological malignancies (comprising patients with B cell or antibody deficiencies) vaccinated with BNT162b2. Here it was observed that only 50% of patients had a BNT162b2-induced T cell response, while this was achieved in 80% of the healthy donors. Thus, the threshold of 80% was chosen, with the aim of providing our study population an immunization comparable to the one achieved in the healthy population vaccinated with the approved vaccines. CoVac-1 induced T cell responses are defined as positive T cell response in Interferon gamm (IFN-γ) ELISPOT assay with spot count at least 2-fold higher than the baseline assay (Visit 1). T cell responses are considered to be positive when the mean spot count per well is at least 3-fold higher than the mean number of spots in the negative control wells (stimulated with a control peptide). Only patients with detectable T cell response to the viral peptide panel ex vivo or after in vitro T cell expansion, and thus general ability to mount an antigen-specific immune response will be considered for the evaluation of sufficient immune responses after one CoVac-1 vaccination. Part II (optional): If there is an insufficient immune response measured by Interferon gamma (IFN-γ) ELISpot in Part I of Phase I on day 28, an additional Part (Part II) of Phase I will start enrollment of 14 subjects receiving two open-label 500 μl subcutaneous injection via needle and syringe of the study IMP (CoVac-1) on day1 and day42.

Phase II (after an amendment to the protocol):

40 subjects will receive an open-label 500 μl subcutaneous injection via needle and syringe of the study IMP (CoVac-1) on d1 and, depending on the data collected in Phase I, a second vaccination on day42 if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years) male or non-pregnant, non-lactating female
2. Primary antibody deficiency syndrome or Secondary antibody deficiency syndrome, defined by one of the following:

   * IgG < 4 g/l
   * Ongoing substitution of immunoglobline for hypogammaglobinemia
   * Anti-CD20 antibody (monospecific) therapy for malignant disease:
   * after combined Anti-CD20 antibody therapy with chemotherapy (e.g. fludarabin, cyclophosphamid, bendamustin, anthracycline, vincristin) or BTK-inhibitors or BCL2-inhibitors (within 1-6 months post therapy)
   * ongoing single agent Anti-CD20 antibody therapy
   * Anti-CD20 antibody maintenance therapy
3. Ability to understand and voluntarily sign an informed consent form
4. Ability to adhere to the study visit schedule and other protocol requirements
5. Female patients of child bearing potential (FCBP) and male patients with partners of child bearing potential, who are sexually active, must agree to the use of two effective forms (at least one highly effective method) of contraception. This should be started from the signing of the informed consent and continue until three months after vaccination. Furthermore, contraception must be carried on by patients receiving B-cell depleting therapies for the whole duration of the treatment.
6. Postmenopausal or evidence of non-child-bearing status. For women of childbearing potential: negative urine or serum pregnancy test within 7 days prior to study treatment. Postmenopausal or evidence of nonchildbearing status is defined as:

   * Amenorrhoea for 1 year or more following cessation of exogenous hormonal treatments
   * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the postmenopausal range for women under 50

Exclusion Criteria:

1. Pregnant or lactating females
2. Participation in any clinical trial with intake of any nonregistered vaccine product
3. Any concomitant disease affecting the effect of the therapeutic vaccine or interfering with the study primary endpoint:

   * Active infection
   * Psychiatric disorders
   * Known systemic anaphylaxis
4. Prior or current infection with SARS-CoV-2 as assessed by medical history and/or by throat/nose swab (PCR) or serologically documented immunization against SARSCoV- 2 (after infection or vaccination)
5. Persisting symptoms developed after SARS-CoV-2 vaccination with an approved vaccine product at study inclusion
6. History of Guillain-Barré syndrome
7. HIV infection, chronic or active hepatitis B or C
8. History of relevant CNS pathology or current relevant CNS pathology (e.g. seizure, paresis, aphasia, cerebrovascular ischemia/haemorrhage, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder, excluding febrile seizures as child)
9. Baseline laboratory CD4+ T cell count < 100 μl
10. The following pre-existing medical conditions:

    * Chronic liver failure defined as Child-Pugh Score ≥B
    * Chronic renal failure defined as GFR <40 ml/min/1,73m2
    * Serious pre-existing cardiovascular disease such as NYHA ≥ III
    * Sickle cell anemia
11. Patients presenting with any clinical, laboratory or radiological signs of tumor-progression
12. Patient receiving active treatment with small molecules, including Tyrosine Kinases-Inhibitors (e.g. Ibrutinib), Proteosome-Inhibitors (e.g. Bortezomib), Bcl-2- Inhibitors (e.g. Venetoclax), Phosphoinositid-3-Kinase- Inhibors (e.g. Idelalisib)
13. Known hypersensitivity to any of the components included in the CoVac-1 vaccine
14. Pre-existing auto-immune disease except for Hashimoto thyroiditis and mild (not requiring immunosuppressive treatment) psoriasis
15. Intention of receiving one dose of an already approved vaccine against SARS-CoV-2 before day 56

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Safety-Vital Signs 1 (Body Temperature) | Day 28
  Body temperature will be measured [temperature in centigrade]
Safety-Vital Signs 2 (Blood Pressure and Pulse) | Day 28
  blood pressure [mmHg] pulse [bpm]
Safety-Eastern Cooperative Oncology Group (ECOG) Status | Day 28
  Scale 0-5, the lower the scale value, the better
Safety-Hematology 1 (Hemoglobin) | day 28
  hemoglobin (Hb). Differential cell counts should be performed at baseline, at each visit during vaccination phase and thereafter at investigators discretion. Clinical status and laboratory parameters are to be followed using individual institutional guidelines and the best clinical judgment of the responsible physician, which can involve more frequent testing.
  Hemoglobin [g/dl ]
Safety-Hematology 2 (White Blood Cells) | day 28
  white blood cells (WBC). Differential cell counts should be performed at baseline, at each visit during vaccination phase and thereafter at investigators discretion. Clinical status and laboratory parameters are to be followed using individual institutional guidelines and the best clinical judgment of the responsible physician, which can involve more frequent testing.
  White Blood Cells [1/µl]
Safety-Hematology 3 (Platelet Count) | day 28
  platelet count (PLT) . Differential cell counts should be performed at baseline, at each visit during vaccination phase and thereafter at investigators discretion. Clinical status and laboratory parameters are to be followed using individual institutional guidelines and the best clinical judgment of the responsible physician, which can involve more frequent testing.
  Platelet Count [1000/µl]
Safety-Hematology 4 (Red Blood Cells) | day 28
  red blood cells (RBC). Differential cell counts should be performed at baseline, at each visit during vaccination phase and thereafter at investigators discretion. Clinical status and laboratory parameters are to be followed using individual institutional guidelines and the best clinical judgment of the responsible physician, which can involve more frequent testing.
  Red Blood Cells [Mio/µl]
T cell response | Day 28
  Blood will be taken before peptide vaccination on V1, and during vaccination phase and follow-up at each visit.
  IFN-gamma ELISPOT Counts

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Salih, Prof. MD, Principal Investigator — University Hospital Tuebingen
Locations (3):
- Germany (3):
  - University Hospital Tuebingen, Tübingen, Baden-Wurttemberg
  - Krankenhaus Nordwest gGmbH Institut für Klinisch-Onkologische Forschung (IKF), Frankfurt am Main, Frankfurt
  - Charité - Universitätsmedizin Berlin Medizinische Klinik m. S. Hämatologie, Onkologie und Tumorimmunologie Charité Campus Benjamin Franklin, Berlin

REFERENCES:
- [Derived] Heitmann JS, Tandler C, Marconato M, Nelde A, Habibzada T, Rittig SM, Tegeler CM, Maringer Y, Jaeger SU, Denk M, Richter M, Oezbek MT, Wiesmuller KH, Bauer J, Rieth J, Wacker M, Schroeder SM, Hoenisch Gravel N, Scheid J, Marklin M, Henrich A, Klimovich B, Clar KL, Lutz M, Holzmayer S, Horber S, Peter A, Meisner C, Fischer I, Loffler MW, Peuker CA, Habringer S, Goetze TO, Jager E, Rammensee HG, Salih HR, Walz JS. Phase I/II trial of a peptide-based COVID-19 T-cell activator in patients with B-cell deficiency. Nat Commun. 2023 Aug 18;14(1):5032. doi: 10.1038/s41467-023-40758-0. PMID 37596280